CLINICAL TRIAL: NCT06162546
Title: ARREST-NEPHROSIS - Austrian Resistant Nephrotic Syndrome Treatment Response Registry and Biobank
Status: Recruiting | Type: Observational
Sponsor: Christoph Aufricht (Other)
Responsible Party: Sponsor-Investigator, Christoph Aufricht, Prof. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: ARREST-NEPHROSIS
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Focal Segmental Glomerulosclerosis; Proteinuria; Nephrotic Syndrome; Nephrotic Syndrome Steroid-Resistant
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria; Nephrotic Syndrome | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARREST NEPHROSIS Participants
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Registry Participation, providing data and clinical specimen

SUMMARY:
Nephrotic syndrome is the clinical phenotype of a heterogeneous group of glomerular diseases that may present with varying degrees of urinary protein loss (proteinuria), dysproteinemia in the blood, fluid retention and impaired renal function.

The AustRian RESistanT NEPHROtic Syndrome Treatment Response RegIStry and Biobank (ARREST-NEPHROSIS) sets out to achieve the following goals, as typical categories of rare disease registries

1. Obtaining real world data on practice patterns and outcomes
2. Networking between affected patients, families, and clinicians.
3. Establish a patient base for facilitated recruitment in studies of drugs, medical devices, and products
4. Development of a Biobank to enable research of potential biomarkers and therapy or disease courses

DETAILED DESCRIPTION:
A significant proportion of patients with nephrotic syndrome remains unresponsive to currently used therapies ("resistant nephrotic syndrome"), the majority of them with focal segmental glomerulosclerosis (FSGS). FSGS is reported as an underlying condition in 5% of adult and 12% of pediatric patients with end-stage kidney disease (ESKD), ultimately requiring renal replacement therapy. The estimated incidence for FSGS is 7 patients per 1 million people.

Despite its clinical and financial burden, the pharmaceutical market for such rare (orphan) diseases is narrow, and industry is less likely to invest in research and to develop treatments for these than for more prevalent medical conditions. However, there remains an urgent need to find new treatments and test their efficacy in suitable trials in resistant nephrotic syndrome.

Patient registries are critical tools to tackle that unmet medical need in orphan diseases. The AustRian RESistanT NEPHROtic Syndrome Treatment Response RegIStry and Biobank (ARREST-NEPHROSIS) therefore sets out to achieve the following goals, in line with typical categories of rare disease registries: (1) networking between affected patients, families, and clinicians; (2) obtaining real world data on practice patterns and outcomes (3); establish a patient base for facilitated recruitment in studies of drugs, medical devices, and products, and (4) development of a biobank to enable research of potential biomarkers predicting disease courses under therapy.

To achieve these goals, the ARREST-NEPHROSIS registry aims for long-term data collection in patients from childhood to adulthood. Patients who fulfill the inclusion criteria (resistance to standard immunosuppressive agents (if clinically indicated, e.g. for primary/non-genetic forms), persistent urinary protein-to-creatinine (UP/C) ratio >1.0 g/g, eGFR > 30 ml/min per 1.73 m2 and a biopsy or a disease-causing genetic mutation associated with nephrotic syndrome) will be invited to the registry, and, after consent, will undergo clinical assessments and receive care as determined by the patient's treating physician. Clinical routine data will be transcribed into the registry to describe patient characteristics (e.g. age, sex, etc.), disease typology (e.g. biopsy and genetics findings, treatment history, etc.), disease activity (e.g. level of proteinuria) and renal function (e.g. eGFR decline).

The continuous prospective assessment of internationally harmonized endpoints suggested by the SONG-GD group (such as proteinuria, including patient reported outcomes (PROs), and the low barrier for access to novel therapeutic studies, will represent an important component of rare disease research in Austria and might ultimately improve health outcomes in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Resistant to standard Immunosuppressive agents (if clinically indicated, e.g. primary/non-genetic forms)
* Persistent urinary protein-to-creatinine (UP/C) ratio >1.0 g/g
* eGFR > 30 ml/min per 1.73 m2
* biopsy or a disease-causing genetic mutation associated with nephrotic syndrome

Exclusion Criteria:

* Inability or unwillingness to comply with repeated assessments
* Objections against participation at discretion of the investigator
* Secondary
* Patients with steroid-dependence/frequently relapsing disease (but achievement of complete remission)

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with nephrotic syndrome are informed about the project as part of a routine check-up and invited to participate by their treating physician. Patients are also informed verbally that there is no obligation to participate and that they can withdraw their willingness to participate at any time.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Obtaining real world data on practice patterns and outcomes in resistant nephrotic syndrome | up to 20 years
Enable networking between patients, families, and clinicians affected by resistant nephrotic syndrome | up to 20 years
Establish a patient base for facilitated recruitment in studies of drugs, medical devices, and products on resistant nephrotic syndrome | up to 20 years
Development of a Biobank to enable research of potential biomarkers and therapy or disease courses | up to 20 years

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Pediatric Nephrology and Gastroenterology, Department of Pediatrics and Adolescent Medicine, Comprehensive Center for Pediatrics, Medical University of Vienna, 1090 Vienna, Austria., Vienna, Austria

IPD SHARING:
Plan to Share IPD: No